CLINICAL TRIAL: NCT06158269
Title: Phase II Clinical Study of Daratumumab Combined With Bortezomib, Lenalidomide and Dexamethasone (DVRd) in the Treatment of Patients With Newly Diagnosed Double-hit Multiple Myeloma
Brief Title: DVRd in the Treatment of Patients With Newly Diagnosed Double-hit Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Qiu Lugui, Prof., Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMY2094
Record Dates: First submitted 2023-09-21; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma
Keywords: double-hit; daratumumab; bortezomib; lenalidomide; minimal residual disease; tailored maintenance therapy
MeSH Terms: conditions — Multiple Myeloma; Neoplasm, Residual

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DVRd group (Experimental): Daratumumab combined with bortezomib, lenalidomide and dexamethasone
  Interventions: Drug: DVRd

INTERVENTIONS:
Drug: DVRd — The patients will receive 4 cycles of DVRd induction therapy. After achieving PR or better response, they will receive stem cell mobilization, collection and the following ASCT. Then, the patients will accept 4 cycles of DVRd consolidation and DVR maintenance therapy. Once they sustain MRD negative condition for at least 12 months, the patients will enter the maintenance stage of lenalidomide monotherapy. Otherwise, the triple drug maintenance therapy will be continued for a total of 24 cycles or until disease progression, death, intolerance, withdrawal due to other reasons, or termination/end of the study.

SUMMARY:
Evaluate the efficacy of DVRd in patients with newly diagnosed double-hit multiple myeloma (MM) and the feasibility of minimal residual disease (MRD) guided maintenance therapy

DETAILED DESCRIPTION:
This study is a single arm phase II study treating patients with newly diagnosed double-hit MM with DVRd induction therapy. This study will enroll 40 patients with double-hit MM who are eligible for autologous stem cell transplantation (ASCT) to evaluate the efficacy of DVRd and the feasibility of MRD guided maintenance therapy. The protocol is: DVRd induction therapy for 4 cycles, followed by ASCT, then DVRd consolidation therapy for 4 cycles, and the last DVR maintenance therapy. After induction therapy, during 60 to 90 days after ASCT, after consolidation therapy, and every 4 cycles during maintenance therapy, the patients will accept MRD monitoring. Patients with MRD negative for at least 12 months will enter the maintenance phase of lenalidomide monotherapy. Otherwise, they will accept DVR maintenance therapy for a total of 24 cycles or until disease progression, death, intolerance, withdrawal due to other reasons, or termination/end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signing the Informed Consent Form (ICF).
2. Age: ≥ 18 years old and < 70 years old.
3. Newly diagnosed MM according to International Myeloma Working Group (IMWG) criteria, with at least one measurable disease: The serum M protein detected by serum protein electrophoresis (SPEP) is ≥ 1g/dL (≥ 10 g/L), or if it is immunoglobulin A (IgA) or immunoglobulin D (IgD) subtype, quantitative levels of total IgA or IgD can be used as a substitute; Or urine M-protein level ≥ 200 mg/24 h; Or if only the serum free light chain (FLC) ratio is abnormal, the affected serum FLC ≥ 100 mg/L (normal FLC ratio: 0.26 to 1.65).
4. At least two high-risk cytogenetic abnormalities: t(4;14), t(14;16), t(14;20), del(17p), gain/amp(1q) (the threshold for copy number variation is 20%, and the threshold for translocation is 10%.
5. The Eastern Cooperative Oncology Group (ECOG) score is 0, 1, or 2 points. The ECOG score of 3 points due to myeloma bone disease can be included.
6. Subjects had not received any anti-MM chemotherapy, extensive pelvic irradiation (more than half of the pelvic area), or anti-MM glucocorticoids, except those who used glucocorticoids for no more than 14 days to control symptoms.
7. Total bilirubin < 1.5 × upper limit of normal (ULN) (total bilirubin in patients with Gilbert's syndrome can be restricted to <3 × ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN.
8. Creatinine clearance rate ≥ 30 mL/min (calculated by cockcroft and Gault formulas).
9. Routine blood test within 7 days before the first day of cycle 1 meets the following criteria: white blood cell (WBC) count ≥ 1.5×10^9/L, absolute neutrophil count ≥ 1.0×10^9/L, hemoglobin ≥ 75 g/L, and platelet count ≥ 75×10^9/L (if bone marrow plasmacytes < 50%) or platelet count ≥ 50×10^9/L (if bone marrow plasmacytes ≥ 50%).
10. Patients receiving erythropoietin, granulocyte colony stimulating factor (G-CSF), granulocyte macrophage colony stimulating factor (GM-CSF), platelet agonists (for example, eltrombopag, thrombopoietin, interleukin-11), must have a 2-week interval between receiving growth factor support and screening assessment.
11. Patients receiving blood product transfusions: at least 2 weeks between hemoglobin assessment and the last red blood cell (RBC) transfusion; at least one week between platelet assessment and the last platelet transfusion.
12. The subjects have no contraindications of receiving prophylactic anticoagulant drug recommended by the study.
13. Female subjects of childbearing age must meet the following two criteria: agree to take effective contraceptive measures from the date of signing the ICF to 3 months after the last administration of the drug; negative serum pregnancy test during screening.

Exclusion Criteria:

1. Primary plasma cell leukemia.
2. Secondary amyloidosis.
3. Central nervous system (CNS) involvement.
4. Patients planning to receive allogeneic hematopoietic stem cell transplantation.
5. Patients with > grade 2 peripheral neuropathy or ≥ grade 2 peripheral neuropathy with pain, regardless of receiving therapy or not.
6. Intolerance, allergy or contraindication to glucocorticoids, bortezomib, lenalidomide or daratumumab.
7. Clinically significant heart diseases: myocardial infarction before screening, or unstable or uncontrollable diseases related to or affecting cardiac function (such as unstable angina, congestive heart failure, New York Heart Association classification III-IV). Uncontrolled arrhythmia or clinically significant electrocardiogram (ECG) abnormalities. During screening, the 12-lead ECG showed a corrected QT interval (QTc) of > 470 msec.
8. Uncontrolled diabetes mellitus and hypertension.
9. Patients with a history of other malignant tumors within 5 years.
10. Active human immunodeficiency virus (HIV) infection or positive serum HIV.
11. Active hepatitis B or C infection. Hepatitis serological test should be performed during screening. If hepatitis B surface antigen (HBsAg) and hepatitis B core antibody (HBcAb) of patients are positive, DNA polymerase chain reaction (PCR) test should be confirmed as negative before enrollment (After anti hepatitis B virus treatment, DNA PCR test should be confirmed as negative before enrollment). If hepatitis C antibody is positive, RNA PCR test should be performed, and the results should be confirmed as negative before enrollment.
12. Pregnant or lactating women.
13. Expected life < 6 months.
14. Any uncontrolled gastrointestinal dysfunction that affects the capacity to ingest or absorb the tablets.
15. A major surgery history within 2 weeks prior to the start of screening, or will not fully recover from the surgery, or are scheduled for surgery during the study period. Kyphoplasty or vertebroplasty is not considered as a major surgery. Notes: Subjects who plan to undergo surgery under local anesthesia can participate in the study.
16. Patients who received attenuated live vaccines within 4 weeks prior to the first administration of the study drug.
17. According to the researcher's judgment, any uncontrolled serious mental illness, physical illness, or other symptoms/conditions that may affect treatment, compliance, or the capacity to sign the ICF.
18. Patients with contraindications to any concomitant drugs or supportive therapy.
19. Patients with any diseases or complications that may interfere with the study procedure.
20. Patients who are unwilling or unable to follow the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
MRD negative rate | through study completion, an average of 3 year
  MRD detected by next generation sequencing

SECONDARY OUTCOMES:
Duration of negative MRD | through study completion, an average of 3 year
  From the first record of negative MRD to the first record of positive MRD or the end of follow-up, whichever came first, assessed up to 3 year
stringent complete response (sCR) | through study completion, an average of 3 year
  stringent complete response
ORR | through study completion, an average of 3 year
  Overall response rate (ORR): Complete response (CR) + Very good partial response (VGPR) + Partial response (PR)
Duration of response (DOR) | through study completion, an average of 3 year
  The duration from the first record of achieving at least PR to the occurrence of progressive disease (PD) or death caused by PD, whichever occurs at first
Mobilization success rate | after all patients accepted stem cell mobilization, an average of 1.5 year
  Mobilization success rate, high-quality mobilization rate and poor-quality mobilization
Progression-free survival (PFS) | through study completion, an average of 3 year
  From date of enrollment of patients until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 year
Overall survival (OS) | through study completion, an average of 3 year
  From date of enrollment of patients until the date of death from any cause, whichever came first, assessed up to 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT06158269/Prot_000.pdf